CLINICAL TRIAL: NCT03427125
Title: A 26-Wk, Phase 3, Open Label (OL) Study With a 12-Wk, Placebo-Controlled, Randomized Withdrawal Period and an OL Safety Extension to Evaluate the Safety and Efficacy of Tenapanor to Treat Hyperphosphatemia in CKD Patients on Dialysis
Brief Title: A Phase 3 Study of Tenapanor to Treat Hyperphosphatemia in ESRD Patients on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TEN-02-301
Record Dates: First submitted 2018-01-19; First posted 2018-02-09 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — tenapanor; Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tenapanor 10 mg, 20 mg, 30 mg BID (Experimental): During the 26-week open label part, all enrolled subjects will receive 30 mg BID doses of tenapanor. Investigators may decrease or increase the dose in 10 mg increments to a minimum of 10 g BIDor a maximum of 30 mg BID
  Interventions: Drug: Tenapanor
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Sevelamer Carbonate (Active Comparator): Subjects randomized into the active control group, for safety analysis, will receive sevelamer carbonate, open label, for the entire 52-week study period. Sevelamer carbonate will be dosed based on package insert instructions (standard of care)
  Interventions: Drug: Sevelamer Carbonate

INTERVENTIONS:
Drug: Tenapanor — Active Drug
  Other Names: RDX5791, AZD1722
  Arms: Tenapanor 10 mg, 20 mg, 30 mg BID
Drug: Placebo — Inactive Drug
  Arms: Placebo
Drug: Sevelamer Carbonate — Active control
  Other Names: Renvela
  Arms: Sevelamer Carbonate

SUMMARY:
This Phase 3, 26-week, open label study with a 12-week, placebo-controlled, randomized withdrawal period followed by an open label long term safety extension will evaluate the safety and efficacy of tenapanor to treat hyperphosphatemia in end-stage renal disease (ESRD) on hemodialysis and peritoneal dialysis.

DETAILED DESCRIPTION:
The study consists of a screening visit, a phosphate binder-free washout period of up to 4 weeks, a 26-week treatment period, an up to 12-week placebo-controlled, randomized withdrawal period, during which patients are randomized 1:1 to either remain on their tenapanor treatment or placebo, followed by an open label safety extension period for a total treatment period of up to 52 weeks. An active control group, for safety analysis only, will receive sevelamer carbonate, open label, for the entire 52-week study period

Depending on increase in serum phosphate (s-P) levels, subjects can be randomized 2 or 3 weeks after being taken off their phosphate lowering medication.

Subjects who qualify to enroll in the study will be randomized 3:1 to either receive tenapanor at a dose of 30 mg bid or sevelamer carbonate.

ELIGIBILITY:
Inclusion Criteria:

* Females must be non-pregnant, non-lactating, and either be post-menopausal for at least 12 months, have documentation of irreversible surgical sterilization, or confirm the use of one of the acceptable contraceptive methods
* Males must agree to avoid fathering a child and agree to use an appropriate method of contraception
* Chronic maintenance hemodialysis 3x a week for at least 3 months
* Chronic maintenance peritoneal dialysis for a minimum of 6 months
* Kt/V ≥ 1.2 at most recent measurement prior to screening
* Prescribed and taking at least 3 doses of phosphate binder per day
* Serum phosphorus levels should be between 4.0 and 8.0 mg/dL at screening
* Unchanged dose of vitamin D or calcimimetics for the last 4 weeks prior to screening
* For enrollment in the study after at least 2 weeks of wash-out, subjects must have serum phosphorus levels of at least 6.0 mg/dL but not more than 10.0 mg/dL and have had an increase of at least 1.5 mg/dL versus pre-wash out value after 2 or 3 weeks wash-out of phosphate binders

Exclusion Criteria:

* Severe hyperphosphatemia defined as serum phosphorus greater than 10.0 mg/dL on phosphate-binders at any time point during clinical routine monitoring for the 3 preceding months before screening visit
* Serum/plasma parathyroid hormone >1200 pg/mL
* Clinical signs of hypovolemia at enrollment
* History of IBD or IBS-D
* Scheduled for living donor kidney transplant, change to peritoneal dialysis, home HD or plans to relocate to another center during the study period
* Positive serology with evidence of significant hepatic impairment or WBC elevation according to the Investigator
* Life expectancy <6 months
* Previous exposure to tenapanor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1559 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, PhD, Study Director — Ardelyx
Locations (2):
- United States (2):
  - Site 529, The Bronx, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Sprague SM, Weiner DE, Tietjen DP, Pergola PE, Fishbane S, Block GA, Silva AL, Fadem SZ, Lynn RI, Fadda G, Pagliaro L, Zhao S, Edelstein S, Spiegel DM, Rosenbaum DP. Tenapanor as Therapy for Hyperphosphatemia in Maintenance Dialysis Patients: Results from the OPTIMIZE Study. Kidney360. 2024 May 1;5(5):732-742. doi: 10.34067/KID.0000000000000387. Epub 2024 Feb 7. PMID 38323855
- [Derived] Silva AL, Chertow GM, Hernandez GT, Lynn RI, Tietjen DP, Rosenbaum DP, Yang Y, Edelstein S. Tenapanor Improves Long-Term Control of Hyperphosphatemia in Patients Receiving Maintenance Dialysis: the NORMALIZE Study. Kidney360. 2023 Nov 1;4(11):1580-1589. doi: 10.34067/KID.0000000000000280. Epub 2023 Oct 19. PMID 37853560
- [Derived] Block GA, Bleyer AJ, Silva AL, Weiner DE, Lynn RI, Yang Y, Rosenbaum DP, Chertow GM. Safety and Efficacy of Tenapanor for Long-term Serum Phosphate Control in Maintenance Dialysis: A 52-Week Randomized Phase 3 Trial (PHREEDOM). Kidney360. 2021 Aug 27;2(10):1600-1610. doi: 10.34067/KID.0002002021. eCollection 2021 Oct 28. PMID 35372979

RESULTS

PARTICIPANT FLOW:
Period: 2 to 4 Week Washout Period
Arm/Group | Tenapanor 10 mg, 20 mg, 30 mg BID | Placebo | Sevelamer Carbonate
Started (All patients were washed off of existing phosphate lowering medication. No patient received study drug during this period) | 0 (No patients received study drug during this period) | 1559 | 0 (No patients received study drug during this period)
Completed | 0 | 564 | 0
Not Completed | 0 | 995 | 0
Not completed — Screen failure (did not meet study entry requirements) | 0 | 995 | 0
Period: 26-Week Treatment Period
Arm/Group | Tenapanor 10 mg, 20 mg, 30 mg BID | Placebo | Sevelamer Carbonate
Started | 423 (Patients were randomized 3:1 to receive tenapanor:sevelamer. The total number of participants receiving tenapanor (423) and sevelamer (141) equal the total number randomized (564).) | 0 (No study participants received placebo during this period) | 141 (Patients were randomized 3:1 to receive tenapanor:sevelamer. The total number of participants receiving tenapanor (423) and sevelamer (141) equal the total number randomized (564).)
Completed | 256 | 0 | 117
Not Completed | 167 | 0 | 24
Period: 12-Week Randomized Withdrawal Period
Arm/Group | Tenapanor 10 mg, 20 mg, 30 mg BID | Placebo | Sevelamer Carbonate
Started | 129 (The 256 participants from the tenapanor group that completed the previous study period were randomized in a double bind manner 1:1 to either stay on tenapanor or placebo.) | 127 (The 256 participants from the tenapanor group that completed the previous study period were randomized in a double bind manner 1:1 to either stay on tenapanor or placebo.) | 117 (Participants that received sevelamer did not participate in this period of the study they continued receiving drug per standard of care.)
Completed | 99 | 99 | 112
Not Completed | 30 | 28 | 5
Period: 14-Week Safety Extension
Arm/Group | Tenapanor 10 mg, 20 mg, 30 mg BID | Placebo | Sevelamer Carbonate
Started | 222 (Participants that dropped out of the previous period due to elevated serum phosphorus could enroll into this safety extension period; that is why the number (222) is higher than the number of participants that completed the previous period) | 0 (There was no placebo group in this period. All participants that received placebo in the previous study period when into the tenapanor group.) | 112
Completed | 205 | 0 | 109
Not Completed | 17 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Placebo was only used in the randomized withdrawal period (RWP). In the RWP, patients from the tenapanor (TEN) group were randomized 1:1 to either remain on TEN or receive a matching placebo. The patients on Sevelamer were not included in this part of the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenapanor 10 mg, 20 mg, 30 mg BID | Placebo | Sevelamer Carbonate | Total
Number analyzed (Participants) | 419 | 0 | 137 | 556
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.74 (12.639) |  | 59.00 (12.638) | 58.05 (12.639)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 |  | 46 | 200
  Male | 265 |  | 91 | 356
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 115 |  | 41 | 156
  Not Hispanic or Latino | 302 |  | 96 | 398
  Unknown or Not Reported | 2 |  | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 |  | 0 | 11
  Asian | 21 |  | 7 | 28
  Native Hawaiian or Other Pacific Islander | 2 |  | 0 | 2
  Black or African American | 195 |  | 60 | 255
  White | 189 |  | 70 | 259
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 1 |  | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.30 (7.505) |  | 31.41 (9.918) | 31.33 (8.159)

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Phosphorus Levels During Placebo Controlled Randomized Withdrawal Period in the Responder Population
Description: Patients with at least a 1.2 mg/dL decrease in serum phosphorus during the first 26 weeks of the study were defined as the responder population.
Time Frame: 12 weeks (randomized withdrawal period)
Population: The sevalmer arm was not included in the randomized withdrawal period. They were treated as an active safety comparator.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tenapanor 10 mg, 20 mg, 30 mg BID | Placebo | Sevelamer Carbonate
Number analyzed (Participants) | 63 | 68 | 0
mg/dL | 0.43 (0.199) | 1.80 (0.196) |
Statistical Analysis 1: Comparison: Tenapanor 10 mg, 20 mg, 30 mg BID vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

2. Secondary Outcome: Change in Serum Phosphorus Levels During Placebo Controlled Randomized Withdrawal Period in the ITT Population
Description: Placebo Adjusted Change in Serum Phosphorus from the beginning to the end of the Randomized Withdrawal Period in all patients
Time Frame: 12 weeks (randomized withdrawal period)
Population: The sevelamer group did not participate in the randomized withdrawal period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tenapanor 10 mg, 20 mg, 30 mg BID | Placebo | Sevelamer Carbonate
Number analyzed (Participants) | 120 | 123 | 0
mg/dL | 0.22 (0.149) | 0.88 (0.150) |
Statistical Analysis 1: Comparison: Tenapanor 10 mg, 20 mg, 30 mg BID vs Placebo; Test type: Superiority; p = 0.0020, ANCOVA

3. Secondary Outcome: Serum Phosphorus From Baseline
Description: Serum Phosphorus from baseline (post washout) to end of 26 week period
Time Frame: 26 weeks (open label treatment period)
Population: There were no placebo during this period and the sevelamer arm was a safety comparator only
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Sevelamer Carbonate: Subjects randomized into the active control group, for safety analysis, will receive sevelamer carbonate, open label, for the entire 52-week study period. Sevelamer carbonate will be dosed based on package insert instructions (standard of care). Serum Phosphorus was not reported.
  Sevelamer Carbonate: Active control
Arm/Group | Tenapanor 10 mg, 20 mg, 30 mg BID | Placebo | Sevelamer Carbonate
Number analyzed (Participants) | 407 | 0 | 0
mg/dL
  Baseline Serum Phosphorus | 7.44 (1.439) |  |
  End of Period serum Phosphorus | 5.88 (1,455) |  |

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tenapanor 10 mg, 20 mg, 30 mg BID | Placebo | Sevelamer Carbonate
All-Cause Mortality (participants affected / at risk) | 12/419 | 1/126 | 5/137
Serious Adverse Events (participants affected / at risk) | 47/419 | 4/126 | 39/137
Other Adverse Events (participants affected / at risk) | 222/419 | 2/126 | 10/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenapanor 10 mg, 20 mg, 30 mg BID (N=419) | Placebo (N=126) | Sevelamer Carbonate (N=137)
pneumonia (Infections and infestations) | 6 (6) | 0 (0) | 8 (8)
Cellulitis (Infections and infestations) | 6 (6) | 1 (1) | 5 (5)
Sepsis (Infections and infestations) | 6 (6) | 1 (1) | 2 (2)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1) | 5 (5)
Fluid Overload (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 6 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 5 (5)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3) | 0 (0) | 7 (7)
Atrial Fibrillation (Cardiac disorders) | 6 (6) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenapanor 10 mg, 20 mg, 30 mg BID (N=419) | Placebo (N=126) | Sevelamer Carbonate (N=137)
Diarrhea (Gastrointestinal disorders) | 222 (222) | 2 (2) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must approve all proposed publications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT03427125/Prot_SAP_000.pdf